CLINICAL TRIAL: NCT03578510
Title: Is the Lower Incidence of Intradialytic Hypotension During Hemocontrol Dialysis in Comparison With Standard Hemodialysis Attributable to Enhanced to Higher Plasma Vasopressin Levels or to Enhanced Sympathetic Activity and/or to Less Nitric Oxide Production
Brief Title: Effect of Plasma Sodium Concentration on Blood Pressure Regulators During Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, dr. C.F.M. Franssen, Principal Investigator, University Medical Center Groningen
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: AVPII study
Record Dates: First submitted 2018-06-12; First posted 2018-07-06 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Patients With End Stage Renal Disease on Hemodialysis
Keywords: Hemodialysis, sodium, endothelium, sympathetic activity, vasopressin
MeSH Terms: conditions — Diabetes Insipidus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHD (Active Comparator): Standard hemodialysis
  Interventions: Device: Hemocontrol hemodialysis; Device: Standard hemodialysis
- HHD (Experimental): Hemocontrol hemodialysis
  Interventions: Device: Hemocontrol hemodialysis; Device: Standard hemodialysis

INTERVENTIONS:
Device: Hemocontrol hemodialysis — Each participating patient underwent one standard hemodialysis and one hemodialysis with Hemocontrol in random order, both 4 hours in total duration. The Hemocontrol system guides the patients' blood volume along a predefined ideal relative blood volume trajectory, by continuously adjusting ultrafiltration volume and dialysate sodium concentration.
Device: Standard hemodialysis — Each participating patient underwent one standard hemodialysis and one hemodialysis with Hemocontrol in random order, both 4 hours in total duration. During standard hemodialysis, a constant ultrafiltration rate and dialysate conductivity was used.

SUMMARY:
Intradialytic hypotension (IDH) is a frequent and serious complication that may occur during hemodialysis treatment. The investigators and others have shown that the Hemocontrol biofeedback system is associated with improved hemodynamic stability. Hemocontrol is a technique that guides the patients' blood volume along a pre-set trajectory by continuously adjusting the ultrafiltration rate and dialysate conductivity. In a recent pilotstudy, the investigators found significantly higher plasma vasopressin levels during the first hour of dialysis with Hemocontrol in comparison with standard hemodialysis. Increased vasopressin levels may contribute to intradialytic hemodynamic stability during hemodialysis by enhanced vasoconstriction. These results, however, did not prove directly that the improved hemodynamic stability with Hemocontrol is indeed caused by higher initial plasma vasopressin levels. Alternative explanations might be that 1) the higher initial plasma sodium levels with Hemocontrol dialysis enhance activity of the sympathetic nervous system directly, causing vasoconstriction and thereby improved hemodynamic stability and/or 2) that the higher initial plasma levels of sodium in Hemocontrol inhibit the release of nitric oxide by the vascular endothelium. Another goal of this study is to investigate whether vasopressin is removed with hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* A thrice-weekly 4 hours hemodialysis schedule
* Dialysis on an arteriovenous fistula
* A usual interdialytic weight gain of ≥2.0 kg

Exclusion Criteria:

* Age<18 years
* Dialysis duration of <4 or >4 hours
* Dialysis frequency of <3 or >3 times a week
* Dialysis on a central venous catheter
* A usual interdialytic weight gain <2 kg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2012-09-17 (Actual); Primary Completion 2013-03-25 (Actual); Study Completion 2013-03-25 (Actual)

PRIMARY OUTCOMES:
Change in plasma vasopressin levels | Before, after 30, 60, 120 and 180 minutes and after dialysis blood is withdrawn from the dialysis line to determine plasma levels of vasopressin.
  Plasma levels of the antidiuretic hormone, i.e. vasopressin

SECONDARY OUTCOMES:
Change in systolic and diastolic blood pressure in mmHg | Before, after 30, 60, 120 and 180 minutes and after dialysis
Change in heart rate in beats per minute | Before, after 30, 60, 120 and 180 minutes and after dialysis
Change in relative blood volume in % | Before, after 30, 60, 120 and 180 minutes and after dialysis
Change in plasma sodium levels in mmol/L | Before, after 30, 60, 120 and 180 minutes and after dialysis

OTHER OUTCOMES:
Change in plasma osmolality levels in milliosmol/kg | Before, after 30, 60, 120 and 180 minutes and after dialysis
Change in nitrite and nitrate levels in µmol/L | Before, after 30, 60, 120 and 180 minutes and after dialysis
Change in plasma noradrenalin levels in mmol/L | Before, after 30, 60, 120 and 180 minutes and after dialysis
Change in heart rate variability in ms | Before, after 30, 60, 120 and 180 minutes and after dialysis
Change in baroreflex sensitivity in ms/mmHg | Before, after 30, 60, 120 and 180 minutes and after dialysis

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ettema EM, Kuipers J, van Faassen M, Groen H, van Roon AM, Lefrandt JD, Westerhuis R, Kema IP, van Goor H, Gansevoort RT, Gaillard CAJM, Franssen CFM. Effect of plasma sodium concentration on blood pressure regulators during hemodialysis: a randomized crossover study. BMC Nephrol. 2018 Aug 22;19(1):214. doi: 10.1186/s12882-018-0997-z. PMID 30134847